CLINICAL TRIAL: NCT04886908
Title: Comparative Retrospective Analysis of Skin Tumors of the Eyelids and Face in 2 Brussels University Hospitals Over 5 Years in Dermatology or Ophthalmology
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Laurence Postelmans, Head of Opthalmology clinic, Brugmann University Hospital
Other Study IDs: CHUB-BOULAKHRIF
Record Dates: First submitted 2021-05-06; First posted 2021-05-14 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data extraction from medical files — Data extraction from medical files

SUMMARY:
Skin cancers are the most common of all cancers. Their incidence has increased sharply over the decades.This increase in incidence partly reflects an aging population and behavioral patterns such as repeated exposure to the sun. Indeed, exposure to UV rays is the predominant factor involved in the pathogenesis of these tumors, hence the fact that they mainly develop in photo-exposed regions such as the cephalic extremity.

The objective of this study is to provide an epidemiological analysis of tumors in the populations of both CHU Brugmann and St Pierre hospitals.

ELIGIBILITY:
Inclusion Criteria:

Final diagnosis confirmed by pathological analysis, epidemiological and clinical information available from patients.

Exclusion Criteria:

Patients who have expressed a refusal to access their medical file or incomplete data will not be taken into account.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Identification of all patients who have undergone surgical excision of benign or malignant facial and/or eyelid tumors over the past 5 years in the Dermatology and/or Ophthalmology Departments of the CHU Saint-Pierre and CHU Brugmann hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Age | 5 minutes
  Age of the patient at the time of diagnose
Sex | 5 minutes
  Sex of the patient
Name of the department in which the patient is followed | 5 minutes
  Ophthalmology-CHU Brugmann hospital or Dermatology-CHU Brugmann hospital or Ophthalmology- CHU St Pierre Hospital or Dermatology-CHU St Pierre Hospital
Tumor anatomical location | 5 minutes
  Eyelids are distributed in their different regions: internal cantus and external cantus, upper eyelid and lower eyelid. Same for the face: ears, zygomatic, forehead, temples, cheeks, nose, upper lip, lower lip, chin, nasolabial fold, preauricular area, retroauricular area, brow bone.
Tumor size | 5 minutes
  Tumor size in millimeters
Laterality | 5 minutes
  Laterality: left, right, median
Multiple or single tumor | 5 minutes
  Multiple or single tumor
Primitive tumor or recidive | 5 minutes
  Primitive tumor or recidive
Risk factor: phototype | 5 minutes
  Phototype 1 to 6 on the Fitzpatrick scale. The Fitzpatrick scale is a numerical classification schema for human skin color. Type 1 is pale skin that always burns, never tans and type 6 is deeply pigmented dark brown to darkest brown skin that never burns.
Risk factor: immunosuppression (yes/no) | 5 minutes
  Pathogenic or iatrogenic, history of malignant skin tumors other than melanoma, personal or family history of melanoma
Risk factor: keratosis | 5 minutes
  Actinic keratosis of the face
Risk factor: solar exposition (yes/no) | 5 minutes
  Lived in a sunny European country> 1 year, lived in a sunny country outside Europe> 1 year, sunbed use> 1 session, history of solar erythema during childhood.
Diagnosis | 5 minutes
  Time between the appearance of the tumor and the first consultation
Locoregional extension report (yes/no) | 5 minutes
  Locoregional extension report (yes/no)
Histological diagnosis of the tumor | 5 minutes
  Histological diagnosis of the tumor
Healthy or invaded margins | 5 minutes
  Healthy or invaded margins
Superficial or infiltrating tumor | 5 minutes
  Superficial or infiltrating tumor
Diagnostic method | 5 minutes
  Diagnostic method: curettage, punch, biopsy, flattening
Surgical management method | 5 minutes
  Biopsy resection, plasty, graft, second-line healing, enucleation, additional treatment: radiotherapy, immunotherapy, liquid nitrogen

CONTACTS AND LOCATIONS:
Overall Officials: Nosria Boulakhrif, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No